CLINICAL TRIAL: NCT03419728
Title: Understanding the Effectiveness of Healthy Families Healthy Futures in Houston, Texas
Brief Title: Federal Evaluation of Selected Programs for Expectant and Parenting Youth
Acronym: PEPY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: The Office of Adolescent Health, HHS (U.S. Federal Agency); Decision Information Resources, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50023
Record Dates: First submitted 2018-01-09; First posted 2018-02-05 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Teen Pregnancy Prevention; Contraceptive Usage
Keywords: Teen pregnancy prevention; Long-acting reversible contraception (LARCs); Healthy Families Healthy Futures; Home visiting
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Families, Healthy Futures (Experimental): Family coaches meet with participating pregnant and parenting females, the woman's partner, and the child. Visit frequency varies from once per week to once per month, depending on the length of time in the program, the client's needs, and the accomplishment of program milestones. In the short term, the program seeks to increase the use of Long-Acting Reversible Contraception (LARC), enhance family functioning including improving father involvement, and to meet the baby's child development needs. In the long term, the program aims to delay subsequent pregnancies, ensure positive child development, and increase parents' self-sufficiency.
  Interventions: Behavioral: Healthy Families, Healthy Futures
- Control group (No Intervention): No active treatment for control group. Control group has access to "business as usual" services in community.

INTERVENTIONS:
Behavioral: Healthy Families, Healthy Futures — Home visiting program for pregnant and parenting teens
  Arms: Healthy Families, Healthy Futures

SUMMARY:
Under contract to the U.S. Department of Health and Human Services (DHHS), Mathematica Policy Research is conducting an impact study of Healthy Families Healthy Futures in Houston, Texas for a Federal Evaluation of Programs for Expectant and Parenting Youth (PEPY). The impact study will be designed to address three main questions:

* Was the program successful in exposing participants to program content, such as information about methods of birth control?
* Was the program successful at improving short-term outcomes, such as use of a LARC and intention to space births?
* To what extent did treatment youth receive the intended program components?

DETAILED DESCRIPTION:
A random assignment design will be used to assess the program's impact on exposure to program content and short term outcomes. Potential study participants were recruited between June 2015 and October 2016, and were considered eligible for participation if they were first time mothers between the ages of 14 and 19, English or Spanish speakers, had not enrolled in the program in the previous six mounts, and were not enrolled in the Nurse Family Partnership program. Potential participants who were eligible and who consented to participate were randomly assigned to (1) a treatment group that was eligible for Healthy Families Healthy Futures (HFHF) services or (2) a control group that was not eligible for HFHF. Random assignment was conducted within two blocks determined by whether study participants were pregnant at the time of random assignment or were parenting at the time of random assignment. The study draws on data from HFHF administrative records on service receipt, a baseline survey administered prior to random assignment, and a follow-up survey administered approximately 12 months after random assignment.

ELIGIBILITY:
Inclusion Criteria:

• Must be expectant or parenting

Exclusion Criteria:

* Participated in HFHF in six months prior to random assignment
* Enrolled in Nurse Family Partnership program at time of random assignment
* Oldest child is older than 3 months at random assignment
* Primary language is neither English nor Spanish

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 248 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Exposure to information on relationships, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas" | 12 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about relationships, dating, or marriage
Exposure to information on parenting, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas" | 12 months
  : Binary variable: equal to one if respondent reported attending a class or session (individual or group) about parenting or how to care for their child
Exposure to information on child healthcare, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas" | 12 months
  Binary variable: equal to one if respondent reported attending a class or session (individual or group) about how to get insurance or apply for Medicaid for their child and where to get health care for their child
Exposure to education related services, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas" | 12 months
  Binary variable: equal to one if respondent reported participating in GED preparation, tutoring, or outside help with school work, or program to prepare for a high school diploma
Exposure to career counseling or job training, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas" | 12 months
  Binary variable: equal to one if respondent reported participating in career counseling or job training
Exposure to information about methods of birth control, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas" | 12 months
  Binary variable: equal to one if respondent reported receiving information from doctor, nurse, home visitor, or clinic regarding methods of birth control
Knowledge of condoms | 12 months
  Continuous variable that is the proportion correct of a mother's responses to six survey items about her knowledge of condoms; each of the six individual item is binary, indicating correct (individual item=1) or incorrect (individual item=0).The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Knowledge of birth control pills | 12 months
  Continuous variable that is the proportion correct of a mother's responses to five survey items about her knowledge of birth control pills; each of the five individual items is binary, indicating correct (individual item=1) or incorrect (individual item=0). The proportion correct ranges from 0 to 1, with higher values indicating great knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Knowledge of IUDs | 12 months
  Continuous variable that is the proportion correct of a mother's responses to six survey items about her knowledge of IUDs; each of the six individual items is binary, indicating correct (individual item=1) or incorrect (individual item=0). The proportion correct can range from 0 to 1, with higher values indicating greater knowledge. Items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Knowledge of other hormonal and LARC methods | 12 months
  Continuous variable that is the proportion correct of a mother's responses to five survey items about her knowledge of other forms of birth control; each of the five individual items is binary, indicating correct (individual item=1) or incorrect (individual item=0) responses. The proportion correct ranges from 0 to 1, with higher values indicating greater knowledge.
Use of a LARC | 12 months
  Binary measure equal to one if the respondent indicated using an IUD or an implant, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Unprotected sex | 12 months
  Binary measure equal to one if the respondent indicated having sexual intercourse in the 3 months prior to the survey and having had sexual intercourse without using birth control, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Intention to space births | 12 months
  Binary variable: equal to one if the woman reports she would like to have her next child two to three years or more than three years from the date of the survey or does not want any more children, and zero if she reports wanting to have her next child less than one year or one to two years from the date of the survey or is pregnant at the time of the survey, as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Mother's engagement in play with child | 12 months
  Multiple-item continuous scale variable that is the average of a mother's responses to five individual categorical survey items; variable ranges from 0 to 3 with higher values indicating more frequent interaction with child. Individual items measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Father's engagement with child | 12 months
  Multiple-item continuous scale variable: average of a mother's responses to eight survey items about her HFHF child's father; variable ranges from 0 to 3 with higher values indicating more frequent interaction with child. Survey items are from the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Quality of co-parenting relationship | 12 months
  Multiple-item continuous scale variable: average of mother's responses to seven survey items; variable ranges from 1 to 5 with higher values indicating a stronger co-parenting relationship. Survey items collected using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Financial support from father | 12 months
  Binary variable: equal to one if mother reports that her child's father covers about half or more of the expenses associated with raising their child and zero if mother reports that her child's father covers less than half of child's costs as measured by the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Capacity for self-sufficiency- Goals, plans, problem solving | 12 months
  Multiple-item continuous scale variable: average of a mother's responses to seven survey items about her goals, focus, and problem solving. Each item ranges from 1 to 4, with higher numbers corresponding to stronger agreement. Items measured using the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Number of well visits | 12 months
  Count variable equal to the respondent's reported number of times in which the child saw a doctor, nurse, or other health care professional for a regular checkup, as reported on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"
Health insurance for child | 12 months
  Binary variable equal to one if the respondent reported having health insurance for her child, as reported on the "Positive Adolescent Futures Final 12 Month Follow-up Survey - Texas"

CONTACTS AND LOCATIONS:
Overall Officials: John Deke, Principal Investigator — Mathematica Policy Research
Locations (1):
- Houston Department of Health; participants' homes, Houston, Texas, United States